CLINICAL TRIAL: NCT02298647
Title: Biomarker for Gangliosidosis: BioGM1 / BioGM2 AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGICAL PROTOCOL
Brief Title: Biomarker for Gangliosidosis: BioGM1/BioGM2 (BioGM1/GM2)
Acronym: BioGM1/BioGM2
Status: Withdrawn | Type: Observational
Why Stopped: Transition to BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BioGM1 / BioGM2
Record Dates: First submitted 2014-10-23; First posted 2014-11-24 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Hepato-splenomegaly; Dysostosis Multiplex; Seizures; Mental Retardation
Keywords: Gangliosidosis; Biomarker
MeSH Terms: conditions — Mucopolysaccharidosis I; Seizures; Intellectual Disability; Gangliosidoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectometry, maximal 10 ml blood will be taken via using a dry blood spot filter card. To proof the cor-rect GM1/GM2 diagnosis in those patients where up to the enrollment into the study no genetic testing has been done, sequencing of GM1/GM2 will be done.
  The analyses will be done at the Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with GM1/GM2-Gangliosidosis or high-grade suspicion for GM1/GM2-Gangliosidosis

SUMMARY:
Development of a new MS-based biomarker for the ear-ly and sensitive diagnosis of GM1/GM2 from blood

DETAILED DESCRIPTION:
Gangliosidosis:

Gangliosides are complex compunds consisting of a glycosphingolipid and a sialic acid and are located at the cell surface where they are responsible for detecting extracellular molecules. Gangliosides are mainly located in the nervous system.

If gangliosides accumulate pathologically throughout the body this is known as Gangliosidosis. There are two main sub-types of Gangliosidosis depending on the deficient enzyme, which are known as GM1 and GM2.

GM1-Gangliosidosis GM1-Gangliosidosis is an autosomal recessive disease. Genetic counselling should be provided to affected families. The disorder is caused by mutations in the GLB1-gene coding for beta-galactosidase. To day, more than 165 mutations have been identified. Deficient enzyme activity leads to toxic accumulation of gangliosides in body tissues, and particularly in the central nervous system (CNS).

The disorder is pan-ethnic, however the worldwide prevalence is not known. Prevalence at birth is estimated to be approximately 1:100,000 to 200,000 live births. High prevalence has been found in Malta and Brazil, and in the Cypriot and Roma populations.

Deficiency of the lysosomal hydrolase, acid β-galactosidase, causes GM1.Three clinical sub-types of GM1-Gangliosidosis are recognized, classified by age of onset, as follows:

* Infantile (type 1): In the most common infantile form, coarse facial features, hepato-splenomegaly, generalized skeletal dysplasia (dysostosis multiplex), macular cherry-red spots, and developmental delay/arrest (followed by progressive neurologic deterioration) usually occur within the first 6 months of life. Nonimmune hydrops fetalis has been reported. An increased incidence of Mongolian spots has also been described. A wide spectrum of variability is observed in the appearance and progression of the typical dysmorphic features. As many as 50% of affected infants have a macular cherry-red spot.
* Juvenile (type 2): The juvenile form is characterized by a later age of onset, less hepatosplenomegaly (if any), fewer cherry-red spots (if any), dysmorphic features, or skeletal changes (vertebral dysplasia may be detected radiographically).
* Adult (type 3): The adult form is characterized by normal early neurologic development, with variable age of clinical presentation. Slowly progressing dementia with parkinsonian features and extrapyramidal disease is common. Intellectual impairment may be initially absent or mild but progresses with time. Generalized dystonia with speech and gait disturbance is the most frequently reported early feature. Typically, no hepato-splenomegaly, cherry-red spots, dysmorphic features, or skeletal changes are present aside from scoliosis (mild vertebral changes may be revealed with radiography), but short stature is common.

GM2-Gangliosidosis The GM2-Gangliosidosis are a group of lysosomal lipid storage disorders caused by mutations in at least 1 of 3 recessive genes: HEXA, HEXB, and GM2A. Normal products of all 3 genes are required for normal catabolism of the GM2 ganglioside substrate. Deficient activity of these enzymes leads to accumulation of the substrate inside neuronal lysosomes, leading to cell death. The products of the 3 genes are, respectively, the alpha subunits of b-hexosaminidase A (Hex A). Hex A is a dimer and has the structure alpha-beta.

β-Hexosaminidase B (Hex B) is a dimer of beta chains. It hydrolyzes GM2 and its neutral asialo derivative GA2. Both subunit precursors acquire the mannose 6-phosphate marker for recognition by lysosomes.

Hexosaminidase S (Hex S) is a dimer of alpha chains; it is a normal constituent of plasma and degrades a wide range of glycoconjugates containing β-linked N-acetylhexosaminyl residues. With lack of beta-subunits the increased polymerization of alpha subunits leads to the in-creased formation of Hex S in Tay - Sachs disease.

GM2A is a cofactor required for the normal function of Hex A; it´s disruption likewise leads to a reduced function of Hex A.

Disease classification:

Tay-Sachs disease Tay-Sachs disease (also known as GM2-Gangliosidosis or hexosaminidase-A deficiency) is an autosomal recessive genetic disorder. In its most common variant (known as infantile Tay-Sachs disease), it causes a progressive deterioration of mental and physical abilities that commences around six months of age and usually results in death by the age of four. The dis-ease occurs when harmful quantities of cell membrane components known as gangliosides accumulate in the brain nerve cells, eventually leading to the premature death of the cells. A ganglioside is a form of sphingolipid, which makes Tay-Sachs-Gangliosidosis a member of the Sphingolipidosis. There is no known cure or treatment.

Tay-Sachs disease is caused by a genetic mutation in the HEXA gene on (human) chromosome 15. A large number of HEXA mutations have been discovered, and new ones are still being reported. These mutations reach significant frequencies in specific populations. French Canadians of south-eastern Quebec have a carrier frequency similar to that seen in Ashkenazi Jews, but carry a different mutation. Cajuns of southern Louisiana carry the same mutation that is seen most commonly in Ashkenazi Jews. HEXA mutations are rare and are most seen in genetically isolated populations. Tay-Sachs can occur from the inheritance of either two simi-lar, or two unrelated, causative mutations in the HEXA gene.

Tay-Sachs disease is classified into several forms, which are differentiated based on the onset age of neurological symptoms.

* Infantile Tay-Sachs disease: Infants with Tay-Sachs disease appear to develop normally for the first six months after birth. Then, as neurons become distended with gangliosides, a relentless deterioration of mental and physical abilities begins. The child becomes blind, deaf, unable to swallow, atrophied, and paralytic. Death usually occurs before the age of four.
* Juvenile Tay-Sachs disease: Juvenile Tay-Sachs disease is rarer than other forms of Tay-Sachs, and usually is initially seen in children between two and ten years old. People with Tay-Sachs disease develop cognitive and motor skill deterioration, dysar-thria, dysphagia, ataxia, and spasticity; they typically die between five and fifteen years old.
* Adult/Late-Onset Tay-Sachs disease: A rare form of this disease, known as Adult-Onset or Late-Onset Tay-Sachs disease usually has its first symptoms during the 30s or 40s. In contrast to the other forms, late-onset Tay-Sachs disease is usually not fatal as the effects can stop progressing. It is frequently misdiagnosed. It is characterized by unsteadiness of gait and progressive neurological deterioration. Symptoms of late-onset Tay-Sachs disease which typically begin to be seen in adolescence or early adulthood - include speech and swallowing difficulties, unsteadiness of gait, spasticity, cognitive decline, and psychiatric illness, particularly a schizophrenia-like psychosis. People with late-onset Tay-Sachs disease frequently become full-time wheelchair users in adulthood.

Until the 1970s and 1980s, when the disease's molecular genetics became known, the juvenile and adult forms of the disease were not always recognized as variants of Tay-Sachs disease. Post-infantile Tay-Sachs was often misdiagnosed as other neurological disorders.

Sandhoff disease Sandhoff disease is a lipid storage disorder characterized by a progressive deterioration of the central nervous system. The clinical symptoms of Sandhoff disease are identical to Tay-Sachs disease. Sandhoff disease is an autosomal recessive genetic disorder caused by an abnormal gene for the beta subunit of the hexosaminidase B enzyme. This gene abnormality results in a deficiency of hexosaminidase A and B that results in accumulation of fats (lipids) called GM2 gangliosides in the neurons and other tissues.

Sandhoff disease, also known as Sandhoff-Jatzkewitz disease, variant 0 of GM2-Gangliosidosis or Hexosaminidase A and B deficiency, is a lysosomal genetic, lipid storage disorder caused by the inherited deficiency to create functional beta-hexosaminidases A and B. These catabolic enzymes are needed to degrade the neuronal membrane components, ganglioside GM2, its derivative GA2, the glycolipid globoside in visceral tissues, and some oligosaccharides. Accumulation of these metabolites leads to a progressive destruction of the central nervous system and eventually to death. The rare autosomal recessive neurodegenera-tive disorder is clinically almost indistinguishable from Tay-Sachs disease, another genetic disorder that disrupts beta-hexosaminidases A and S.

There are three different types of Sandhoff disease, classic infantile, juvenile, and adult late onset. Each form is classified by the severity of the symptoms as well as the age in which the patient shows these symptoms:

* Classic infantile form: Classic infantile form of the disease is classified by the development of symptoms anywhere from 2 months to 9 months of age. It is the most severe of all of the forms and will lead to death before the patient reaches the age of three. This is the most common and severe form of Sandoff disease. Infants with this disorder typically appear normal until the age of 3 to 6 months, when development slows and muscles used for movement weaken. Affected infants lose motor skills such as turning over, sitting, and crawling. As the disease progresses, infants develop seizures, vision and hearing loss, mental retardation, and paralysis. An eye abnormality called a cherry-red spot, which can be identified with an eye examination, is characteristic of this disorder. Some infants with Sandhoff disease may also have enlarged organs (or-ganomegalie) or bone abnormalities. Children with the severe form of this disorder usually live only into early childhood.
* Juvenile form: Juvenile form of the disease shows symptoms starting at age 3 ranging to age 10 and although the child usually dies by the time they are 15, it is possible for them to live longer if they are under constant care.
* Adult onset form: Adult onset form of the disease is classified by its occurrence in older individuals and has an effect on the motor function of these individuals and it is not yet known if Sandhoff Disease will cause these individuals to have a decrease in their life span.

Both Juvenile and Adult onset forms of Sandhoff disease are very rare. Signs and symptoms can begin in childhood, adolescence, or adulthood and are usually milder than those seen with the infantile form of Sandhoff disease. As in the infantile form, mental abilities and coordination are affected. Characteristic features include muscle weakness, loss of muscle coordination (ataxia) and other problems with movement, speech problems, and mental illness. These signs and symptoms vary widely among people with late-onset forms of Sandhoff disease.

Sandhoff disease symptoms are clinically indeterminable from Tay-Sachs disease. The classic infantile form of the disease has the most severe symptoms and is incredibly hard to diagnose at this early age. The first signs of symptoms begin before 6 months of age and the parents' notice when the child begins digressing in their development. If the children had the ability to sit up by themselves or crawl they will lose this ability. This is caused by a slow deterioration of the muscles in the child's body from the build-up of GM2 gangliosides. Since the body is unable to create the enzymes it needs within the central nervous system, it is unable to attach to these gangliosides to break them apart and make them non-toxic. With this build-up there are several symptoms that begin to appear such as muscle/motor weakness, sharp reaction to loud noises, blindness, deafness, inability to react to stimulants, respiratory problems and infections, mental retardation, seizures, cherry red spots in the retina, enlarged liver and spleen (hepatosplenomegaly), pneumonia, or bronchopneumonia.

The other two forms of Sandhoff disease have similar symptoms but to a lesser extent. Adult and juvenile forms of Sandhoff disease are rarer then the infantile form. In these cases victims suffer cognitive impairment (retardation) and a loss of muscle coordination that impairs and eventually destroys their ability to walk; the characteristic red spots in the retina also develop. The adult form of the disease, however, is sometimes milder, and may only lead to muscle weakness that impairs walking or the ability to get out of bed.

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to validate this new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

* Informed consent will be obtained from the parents before any study related procedures.
* Patients of both genders aged 2 months and older
* The patient has a diagnosis of GM1/GM2-Gangliosidosis or a high-grade suspicion for GM1/GM2-Gangliosidosis
* High-grade suspicion for GM1 or GM2 present, if one or more inclusion criteria are valid:

Positive family anamnesis for GM1 or GM2 disease

Neurodegenerative symptoms

Skeletal symptoms

Cherry Red Spot

EXCLUSION CRITERIA:

* No Informed consent from the parents before any study related procedures.
* No diagnosis of GM1/GM2 disease or no valid criteria for profound suspicion of GM1/GM2 -disease
* Patients of both genders younger than 2 months

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with GM1/GM2-Gangliosidosis or high-grade suspicion for GM1/GM2-Gangliosidosis
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagnosis of GM1/GM2-Gangliosidosis from blood | 24 months
  New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

SECONDARY OUTCOMES:
Testing for clinical robustness, specificity and long-term stability of the biomarker | 36 months
  the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (5):
- Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt
- Centogene AG, Rostock, Germany
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided